CLINICAL TRIAL: NCT03979014
Title: Nonavalent Prophylactic HPV Vaccine (GARDASIL9) After Local Conservative Treatment for Cervical Intra-epithelial Neoplasia: a Randomised Controlled Trial - The NOVEL Trial
Brief Title: Nonavalent Prophylactic HPV Vaccine (GARDASIL9) After Local Conservative The NOVEL Trial
Acronym: NOVEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C/39/2018
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Neoplasia
Keywords: Neoplasia; Cervix cancer; Vaccination; Coloscopy
MeSH Terms: conditions — Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The patients and clinicians will not be blinded but the laboratory staff performing the HPV assays on vaccinated and non-vaccinated arms will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccinated Arm (Experimental): Add Vaccine
  Interventions: Biological: Gardasill 9™ vaccine
- Control (No Intervention): No intervention

INTERVENTIONS:
Biological: Gardasill 9™ vaccine — 3 doses of Gardasill 9™ vaccine 0.5 ml administered 3 times at 0, 2 and 6 month
  Arms: Vaccinated Arm

SUMMARY:
The researchers involved in this new study are interested in whether giving a HPV vaccine to women at the same time as conisation can lead to a greater rate of HPV clearance compared to conisation on its own, and a result reduce the occurrence of further infection and high grade CIN. The study will do this by using a specific HPV vaccine called Gardasil 9™ which protects against 9 types of HPV infection (types 6, 11, 16, 18, 31, 33, 45, 52 and 58).

DETAILED DESCRIPTION:
The human papilloma virus (HPV) can cause high grade intra-epithelial neoplasia (CIN) in women, a condition where there are abnormal cells on the surface of the cervix (the opening to the vagina from the womb). High grade CIN can develop into cervical cancer, and standard treatment is a surgical procedure called conisation, where a scalpel or laser is used to remove a cone-shaped piece of the cervix containing the abnormal cells. HPV vaccines are routinely used in adolescent girls as part screening programmes to prevent cervical cancer (12-18 years of age in the UK).

The NOVEL study will compare the vaccine approach with standard treatment in a randomised controlled trial, where eligible women will be randomly allocated to one of the following:

Arm 1: Local Cervical treatment and vaccination with Gardasil 9, followed by additional vaccinations 2 and 6 months after conisation Arm 2: Local Cervical Treatment and Observation

This study is for women aged 18-55 years of age with biopsy confirmed high-grade CIN. 1000 women will be recruited at colposcopy clinics in the UK, Finland and Sweden. Women will be followed up for a maximum of two and a half years.

ELIGIBILITY:
Inclusion Criteria

Patients who meet all of the following inclusion criteria will be considered eligible for this study:

1. Female (18-55y) attending for local treatment for presumed CIN2 (cytological and colposcopy impression) OR presumed CIN3 (cytological and colposcopy impression) OR presumed cGIN/AIS (cytological and colposcopy impression) OR biopsy-confirmed CIN2 OR biopsy-confirmed CIN3 OR biopsy-confirmed CGIN/AIS
2. Written informed consent obtained from the subject prior to enrolment
3. Free of other relevant health problems as established by medical history and clinical examination, e.g. immunosuppression
4. Patients who the investigator believes can and will comply with the protocol requirements (e.g. attendance at clinic appointments and return for follow-up visits)

Exclusion criteria

Patients who meet any of the following exclusion criteria will not be eligible for this study:

1. Use of other investigational/non-registered product within 30 days preceding the 1st vaccine dose
2. Continuous administration of immunosuppressants
3. Previous vaccination against HPV
4. Cancer or autoimmune disease under treatment. Patients who have a history of cancer or autoimmune disease but are not currently being treated for the condition will be included
5. Any confirmed or suspected immunosuppressive condition, including HIV infection
6. History of allergic disease or any neurologic disorders likely to interact with study vaccination
7. Acute febrile disease at enrolment (will be postponed)
8. Pregnant women or women intending to get pregnant during the next 6 months (if pregnant during follow-up, remaining doses will be delayed until after delivery)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1099 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Incidence of HPV infection in women with high grade cervical intra-epithelial neoplasia after vaccine Gardasil 9™ assess by laboratory test | 2 years after first dose of vaccine
  High grade CIN is a condition where there are abnormal cells on at least two-thirds of the surface of the cervix (the opening to the vagina from the womb). Gardasil 9™ will be given at the same time as localised cervical treatment, a procedure which uses a scalpel or laser to remove a cone-shaped piece of the cervix containing the area with abnormal cells.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kyrgiou, MBBS, FRCP, Principal Investigator — Imperial College London
Locations (13):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere
- Sweden (3):
  - Regionhälsan Masthugget Clinic of Obstetrics and Gynecology, Gothenburg
  - Sahlgrenska University Hospital, Gothenburg
  - Frölunda Specialist Hospital Gynecology Clinic, Västra Frölunda
- United Kingdom (8):
  - St James's University Hospital, Leeds, Leeds, England
  - Guy's and St Thomas' NHS Foundation Trust, London, England
  - West Middlesex University Hospital, London, England
  - St. Mary's Hospital - Manchester University NHS Foundation Trust, Manchester, England
  - Whittington Health NHS Trust, Middlesex, England
  - Nottingham University Hospitals NHS Trust, Nottingham, England
  - Royal Preston Hospital - Lancashire Teaching Hospitals NHS Trust, Fulwood, Preston
  - St Mary's Hospital - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joura E, Kjaer SK, Bautista O, Luxembourg A, Saah A, Giuliano A. Effect of Prior 9-Valent Human Papillomavirus Vaccination on Subsequent Lower Genital Tract Dysplasia After Cervical Excisional Surgery. Obstet Gynecol. 2026 Jan 1;147(1):73-82. doi: 10.1097/AOG.0000000000006113. Epub 2025 Oct 30. PMID 41166720